CLINICAL TRIAL: NCT03208101
Title: A Single-center, Randomized, Active-controlled, Parallel-group, Open-label, Phase I Study to Evaluate Safety and Immunogenicity of Single Injection of LBVD or Eupenta Co-administered With Imovax Polio in Healthy Adults
Brief Title: A Study to Compare LBVD to Eupenta and Imovax Polio in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VDCL001
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2018-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B; Haemophilus Influenzae Type b Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): DTP-HepB-IPV-Hib vaccine
  Interventions: Biological: DTP-HepB-IPV-Hib vaccine
- Control group (Active Comparator): DTP-HepB-Hib vaccine & IPV
  Interventions: Biological: DTP-HepB-Hib vaccine & IPV

INTERVENTIONS:
Biological: DTP-HepB-IPV-Hib vaccine — Hexavalent vaccine (DTP-HepB-IPV-Hib vaccine: Diphtheria-Tetanus-Pertussis-Hepatitis B-Inactivated Poliovirus-Haemophilus influenzae type b vaccine)
  Arms: Test group
Biological: DTP-HepB-Hib vaccine & IPV — Pentavalent vaccine (DTP-HepB-Hib vaccine: Diphtheria-Tetanus-Pertussis-Hepatitis B-Haemophilus influenzae type b vaccine)+ IPV(Inactivated poliovirus vaccine)
  Arms: Control group

SUMMARY:
This is a single-center, randomized, active-controlled, parallel-group, open-label, phase I study to evaluate safety and immunogenicity of single injection of LBVD or Eupenta co-administered with Imovax Polio in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 19 and 55 years of age at the time of Visit 1 (Screening)
2. Persons who or whose legal representatives have voluntarily signed an informed consent after receiving explanation about the objectives, methods, effects, etc. of the clinical study
3. Persons who are surgically sterile, postmenopausal women, or agree to use contraceptive measures

Exclusion Criteria:

1. Persons who have an experience of participation in another interventional clinical study within 3 months prior to Visit 1 (Screening)
2. Persons who have a record of vaccination with the tetanus toxoid (TT)/tetanus diphtheria (Td)/tetanus diphtheria pertussis (Tdap) vaccine or other vaccines containing tetanus-diphtheria for adults or who are suspected to have been vaccinated with either of them within 5 years prior to Visit 1 (Screening)
3. Persons who were vaccinated within 4 weeks prior to Visit 1 (Screening) or who are scheduled to be vaccinated with the vaccines other than the study vaccine during the study period
4. Persons with a history of diphtheria, tetanus, pertussis, hepatitis B virus, polio virus, or the invasive diseases caused by Haemophilus influenzae type b

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with immediate reactions | For 30 minutes after the vaccination
  Immediate reactions after vaccination with the study vaccine mean all the signs and symptoms occurring within 30 minutes after the vaccination.
Number of subjects with solicited adverse events | For 14 days after the vaccination [Day 1-15]
  Solicited adverse events are classified into the local(pain, tenderness, erythema/redness, induration/swelling) and systemic(fever, fatigue, chills/shivering, myalgia, headache, arthralgia, decreased appetitie, diarrhea, nausea/vomiting, rash) signs and symptoms.
Number of subjects with any unsolicited adverse events | For 28 days (+7 days of window period) after the vaccination [Day 1-29]
  Unsolicited adverse events mean all the adverse events excluding the immediate reactions after vaccination with the study vaccine and the solicited adverse events.

SECONDARY OUTCOMES:
Proportions of the subjects who have shown seroprotection/vaccine-response to each antigen and the subjects who have shown seroconversion 28 days post-vaccination with the study vaccine (Day 29) compared to pre-vaccination. | Day 29 (+7 days window period)
  Immunogenicity of each components (antibodies against Diphtheria, Tetanus, Pertussis, Polio, Hepatitis B, and Haemophilus influenzae type b
GMC or GMT values for each antigen prior to and 28 days post-vaccination with the study vaccine (Day 29) | Day 29 (+7 days window period)
  Immunogenicity of each components (antibodies against Diphtheria, Tetanus, Pertussis, Polio, Hepatitis B, and Haemophilus influenzae type b

CONTACTS AND LOCATIONS:
Overall Officials: WJ Kim, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No